CLINICAL TRIAL: NCT07039617
Title: A Randomized Parallel Clinical Trial of AIDANET, an Automated Insulin Delivery Algorithm, in Fully Closed-Loop Vs Hybrid Closed-Loop Mode In Adults With Type 1 Diabetes
Brief Title: AIDANET At Home Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sue Brown (Other)
Collaborators: Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Sue Brown, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 302656; 5R01DK129553 (NIH)
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
Keywords: Automated Insulin Delivery (AID); Fully Closed Loop (FCL); Hybrid Closed Loop (HCL); Specifically modified Mobi System; Automated Insulin Delivery as Adaptive NETwork (AIDANET)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A (Experimental): Group A: AID first followed by AIDANET-FCL, AIDANET-HCL and then AIDANET-FCL-HCL mix
  Interventions: Device: AIDANET + FCL; Device: AIDANET + HCL; Device: AIDANET in FCL-HCL-mixed mode; Other: Automated Insulin Delivery (AID) (usual care)
- Group B (Experimental): Group B: AIDANET-FCL first followed by AIDANET-HCL, AIDANET- FCL-HCL mix and AID
  Interventions: Device: AIDANET + FCL; Device: AIDANET + HCL; Device: AIDANET in FCL-HCL-mixed mode; Other: Automated Insulin Delivery (AID) (usual care)

INTERVENTIONS:
Device: AIDANET + FCL — All participants will use AIDANET in fully closed loop (FCL) mode with instructions to avoid announcing meal boluses whenever possible during the four weeks.
Device: AIDANET + HCL — All participants will use AIDANET in hybrid closed loop (HCL) mode with instructions to announce all meal boluses using carbohydrate counting or easy bolus during the four weeks. All components of AIDANET will remain active during this phase but BPS in particular is expected to be triggered less often due to meal announcements.
Device: AIDANET in FCL-HCL-mixed mode — All participants will use AIDANET with instructions to choose whether to use fully closed loop (FCL) or hybrid closed loop (HCL) mode with meal announcements (carb counting or easy bolus) per their discretion each day.
Other: Automated Insulin Delivery (AID) (usual care) — Participants will manage their diabetes as they normally do at home.

SUMMARY:
A randomized cross-over trial assessing glycemic control on Automated insulin delivery as Adaptive Network (AIDANET) algorithm when used in three modes: AIDANET-Fully Closed Loop (FCL), AIDANET-Hybrid Closed Loop (HCL) and AIDANET allowing a mix between FCL and HCL. There will be an Automated Insulin Delivery (AID) phase with participants using their home devices and/or study continuous glucose monitor (CGM) and study-provided commercial Mobi system without AIDANET.

DETAILED DESCRIPTION:
This study is a randomized cross-over trial comparing AIDANET used in three different modalities to currently available AID systems (usual care). For two 4-week phases the participants will first use the system in predetermined modality (HCL or FCL) in random order. The AIDANET system is designed to work both in full closed loop (no meal information) and in hybrid closed-loop, with carbohydrate announcement (standard bolus calculator) or easy bolus (announce timing but not carbohydrate amount), as requested by the user. During a third 4-week long phase, all participants will continue to use the system as befits their preferences (no modality will be imposed, and the user is free to go back and forth between modalities). In addition, the participant will spend 4 weeks using a usual care AID system either before the first AIDANET phase (randomization Group A) or after the last AIDANET phase (randomization Group B).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of Type 1 Diabetes for at least one year.
3. Having used an Food and Drug Administration (FDA) approved AID system within the last six months (can be intermittent use).
4. Currently using insulin for at least six months.
5. Willingness to switch to use an FDA-approved personal insulin for the study pump (e.g., lispro or aspart, or biosimilar FDA-approved products) as directed by the study team.
6. Has one or more supportive companions knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff who either lives with participant or located within approximately 30 minutes of participant and able to locate participant in the event of an emergency.
7. Participant not currently known to be pregnant or breastfeeding.
8. If participant capable of becoming pregnant, must agree to use a form of contraception to prevent pregnancy while a participant in the study (e.g. hormonal contraception, abstinence from heterosexual intercourse). A negative serum or urine pregnancy test will be required for all participants of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
9. Willingness to wear a Dexcom CGM during each of the four study phases.
10. Willingness to use the study AIDANET system (CGM, pump, and phone) during the relevant study periods.
11. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial.
12. Willingness to participate in all study procedures including in person training.
13. Access to internet at home and willingness to upload data during the study as needed.
14. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol.
15. Participant is proficient in reading and verbal communication in English.

Exclusion Criteria:

1. Plans to start a new non-insulin glucose-lowering agent (e.g. glucagon-like peptide-1 (GLP-1) receptor agonists, Symlin, (DPP-4 inhibitors, also known as dipeptidyl peptidase 4). Participants may be on a stable dose of such an agent for at least the past month.
2. Current use of sulfonylurea medications.
3. Current use of an Sodium-Glucose Cotransporter 2 (also known as a SGLT-2 or SGLT-1/2 inhibitor) due to risk of euglycemic diabetic ketoacidosis (DKA).
4. Hemophilia or any other bleeding disorder.
5. History of severe hypoglycemic events with seizure or loss of consciousness in the last 12 months.
6. History of DKA event in the last 12 months.
7. Currently on peritoneal or hemodialysis.
8. Currently being treated for adrenal insufficiency.
9. Currently being treated for a seizure disorder.
10. Hypothyroidism or hyperthyroidism is not adequately treated.
11. Use of oral or injectable steroids at the time of enrollment.
12. Known ongoing adhesive intolerance that is not well managed.
13. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk.
14. Participation in another interventional trial at the time of enrollment.
15. Participant with a direct supervisor at work/school who is involved in the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Time in Range (70-180 mg/dL) | 16 weeks
  * Computed as the number of estimated glucose values ≥70mg/dL and <180mg/dL divided by the number of valid values (defined as a number between 39 and 401)
  * Outcome is computed if:
    * >4032 values are recorded (availability condition, 2 weeks equivalent)
    * AND there is >70% values between the first recorded EGV of the analysis window and the last (density condition)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals in the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after the publication of the manuscript.
Access Criteria: The Data Sharing Agreements will be formulated by the study team